CLINICAL TRIAL: NCT02746783
Title: Immunogenicity (Humoral and Cellular Immune Responses) and Safety of the Seasonal Flu Vaccine in Elderly and in SOT Recipients
Brief Title: Immunogenicity and Safety of the Seasonal Flu Vaccine in Elderly and in SOT Recipients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Giuseppe Pantaleo, Prof. Giuseppe Pantaleo, University of Lausanne Hospitals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Vaccinâge 2013-15
Record Dates: First submitted 2014-08-08; First posted 2016-04-21 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Active Comparator): Single dose of MUTAGRIP® containing A/California/7/2009 (H1N1); A/Texas/50/2012 (H3N2); B/Massachusetts/2/2012.
  Interventions: Drug: Single dose MUTAGRIP® influenza vaccine
- Group 2 (Experimental): Double dose of MUTAGRIP® (one dose into the right deltoid area and the other one into the left deltoid area) containing A/California/7/2009 (H1N1); A/Texas/50/2012 (H3N2); B/Massachusetts/2/2012.
  Interventions: Drug: Double dose of MUTAGRIP® influenza vaccine

INTERVENTIONS:
Drug: Single dose MUTAGRIP® influenza vaccine — All subjects will receive either a single or double doses of MUTAGRIP® containing A/California/7/2009 (H1N1); A/Texas/50/2012 (H3N2); B/Massachusetts/2/2012. The double dose regimen will be administered at the same time.
  Arms: Group 1
Drug: Double dose of MUTAGRIP® influenza vaccine — All subjects will receive either a single or double doses of MUTAGRIP® containing A/California/7/2009 (H1N1); A/Texas/50/2012 (H3N2); B/Massachusetts/2/2012. The double dose regimen will be administered at the same time.
  Arms: Group 2

SUMMARY:
This study will assess the effect of a different dose of the seasonal flu vaccine 2013-2015 on the immune response to improve the investigators understanding of cellular and humoral immune responses induced. The scope of this study is to determine the profile of cellular activation and antibody production in the ageing immune system following flu immunization.

This study will enroll 100 male or female subjects ≥65 year old and 90 transplant recipients. These persons will be deemed to be " at risk " in case of influenza infection and should be vaccinated according to Swiss Federal Office of Public Health. A medical doctor from the CHUV will inform the patients about the present study and ask them whether they would be willing to participate in the study.

All subjects will be distributed between the two groups according to a computer-generated randomization sequence. The randomization will be done in blocks to ensure balance across groups. The participants and site staff will not be blinded due to the different administration assignments.

Group 1 subjects will receive a single dose and group 2 subjects a double dose of MUTAGRIP® manufactured by Sanofi Pasteur containing A/California/7/2009 (H1N1); A/Texas/50/2012 (H3N2); B/Massachusetts/2/2012. Vaccine immunogenicity and safety will be assessed 1, 2, 4 and 24 weeks after vaccination.

Study duration per volunteer is 6 months after vaccination.

ELIGIBILITY:
Elderly:

Inclusion Criteria:

* Age ≥65 year old.
* Able to give informed consent.
* Necessity to receive influenza seasonal vaccination in 2013-2015.
* Availability for the duration of the study and willingness to attend all scheduled visits.
* Hemoglobin value ≥100 g/l , Leukocytes ≥3.5 G/L, Platelets count ≥100 G/l at the time of screening, or determined within 8 weeks before screening in the course of regular medical examination and validated by the medical doctor.

Solid-organ transplant recipients Inclusion criteria Age ≥18 year old Solid organ transplantation >3 months before vaccination Stable patient followed at the outpatient clinic of the Transplantation Center Able to give informed consent. Necessity to receive influenza seasonal vaccination. Availability for the duration of the study and willingness to attend all scheduled visits.

Exclusion criteria Previous life-threatening reaction to influenza vaccine (i.e. Guillain-Barre Syndrome) Ongoing therapy for rejection Febrile illness in the past two weeks

Exclusion Criteria:

* Contraindication against seasonal flu vaccination.
* Use of any investigational or non-registered drug or vaccine within 30 days preceding the first dose of the study vaccine, or planned use during the study period and safety follow-up.
* Immunodeficiency or chronic administration (defined as more than 14 consecutive days) of immunosuppressive or other immune-modifying drugs within six months prior to the first vaccine dose. (For corticosteroids, this will mean prednisone, or equivalent, ≥0.5 mg/kg/day. Inhaled and topical steroids are allowed).
* Hypersensitivity to the active substances, to any of the excipients, to eggs, chicken proteins, neomycin, formaldehyde and octoxinol 9.
* Acute disease at the time of enrollment [Acute disease is defined as the presence of a moderate or severe illness with or without fever. All vaccines can be administered to persons with a minor illness such as diarrhea, mild upper respiratory infection with or without low-grade febrile illness, i.e., temperature <38°C].
* An unstable chronic condition (unstable chronic renal failure, unstable diabetes, unstable chronic cardiac condition, uncontrolled asthma, etc.).
* Receipt of blood-derived products (immunoglobulin; plasma) within 120 days prior to enrollment.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 163 (Actual)
Dates: Start 2013-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Immunogenicity | weeks 2, 4 and 24 after vaccination
  Humoral immune responses (antibodies directed against all three strains A/California/7/2009 (H1N1); A/Texas/50/2012 (H3N2); B/Massachusetts/2/2012).
Change from Baseline in Immunogenicity | weeks 1, 2, 4 and 24 after vaccination
  Cellular immune responses directed against all three strains A/California/7/2009 (H1N1); A/Texas/50/2012 (H3N2); B/Massachusetts/2/2012.

SECONDARY OUTCOMES:
Number of Adverse Events as a Measure of Safety and Tolerability | 24 weeks after vaccination
  To evaluate safety and tolerability of the influenza vaccine (split virion, inactivated), MUTAGRIP®, administered in single or double dose.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Pantaleo, Prof., Principal Investigator — Vaccine and Immunotherapy Center (VIC) of the Centre Hospitalier Universitaire Vaudois (CHUV), Switzerland
Locations (1):
- Vaccine and Immunotherapy Center (VIC) of the Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Mombelli M, Rettby N, Perreau M, Pascual M, Pantaleo G, Manuel O. Immunogenicity and safety of double versus standard dose of the seasonal influenza vaccine in solid-organ transplant recipients: A randomized controlled trial. Vaccine. 2018 Oct 1;36(41):6163-6169. doi: 10.1016/j.vaccine.2018.08.057. Epub 2018 Sep 1. PMID 30181045